CLINICAL TRIAL: NCT05467501
Title: Principal Investigator
Brief Title: Effect of Therapeutic Ultrasound Versus Anti-inflammatory Drugs in the Treatment of Trigger Finger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eslam Elsayed Ali Shohda (Other Government)
Responsible Party: Sponsor-Investigator, Eslam Elsayed Ali Shohda, Dr, General Committee of Teaching Hospitals and Institutes, Egypt
Organization: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GeneralCTHI
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Trigger Finger
Keywords: Trigger Finger; Therapeutic Ultrasound
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Masking Description: Patients will not know the actual ultrasound application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): Therapeutic ultrasound application. US parameters are 0.8 W/cm for intensity, 3 MHz for frequency and 5 min application. The device that will be used is medserve, England (the head of the device is 5cm). The physical therapy will by 6 sessions (every day). PT sessions will be done by the same physical therapist.
  Interventions: Device: Theraputic ultrasound
- placepo group (Active Comparator): group B will have a non-steroidal anti-inflammatory drug as prescribed by the same orthopedist and 2 session of massage with the head of ultrasound.
  Interventions: Device: Theraputic ultrasound

INTERVENTIONS:
Device: Theraputic ultrasound — Therapeutic ultrasound
  Other Names: antiinflamatory drug

SUMMARY:
to determine the effect of US on pain intensity in TF patients 2) to determine the effect of US on number of daily finger triggering in TF patients.

DETAILED DESCRIPTION:
Trigger finger (T.F) is a disorder characterized by snapping or locking of a finger. Painful popping or clicking sound is elicited by flexion and extension of the involved digit . It is a multifactorial disease. The common mechanism of triggering is that there is a mismatch of diameter between flexors tendons and the annular pulley (retinacular sheath) of the finger. Some studies found inflammatory cells as a part of the pathology, hence anti-inflammatory drugs are the first line of treatment .

Therapeutic ultrasound (US) is a form of acoustic energy which is often used in physical therapy. When US enters the body, it can affect the cells and tissues through thermal and non-thermal mechanisms. While a thermal mechanism has a direct heating effect which promotes anti-inflammatory response with increase blood flow, evidence indicates, however, that non thermal mechanisms are thought to play a primary role in producing a therapeutically significant biological effect (i.e. the stimulation of tissue regeneration) . So my question is in T.F patients does therapeutic ultrasound decrease pain more than anti-inflammatory drugs?

ELIGIBILITY:
Inclusion Criteria:

1 - patients will be included to this study if they are trigger finger patients ( clinically evaluated and refereed by orthopedist).

Exclusion Criteria:

1 - complete locked finger. 2-Ages below 18 y. 3-Patients with any other hand pathology .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 6 month - 1 year
  measured by visual analog scale

SECONDARY OUTCOMES:
number of daily finger triggering | 6 month - 1 year

IPD SHARING:
Plan to Share IPD: Undecided
to think about important or not